CLINICAL TRIAL: NCT07265856
Title: The Effect of a Comprehensive Dementia Education Program on Improving Attitudes Toward People Living With Dementia: a Randomized Controlled Trial
Brief Title: The Effect of a Comprehensive Dementia Education Program on Improving Attitudes Toward People Living With Dementia
Acronym: VReducationRCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Airlangga (Other)
Collaborators: Chiba University (Other)
Responsible Party: Principal Investigator, Dianis Wulan Sari, Principal Investigator, Universitas Airlangga
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3922-KEPK; 39922-KEPK (Other: Universitas Airlangga)
Record Dates: First submitted 2025-11-16; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Dementia
Keywords: Aged; Dementia; Education program; Healthcare student; Long-term care; Virtual reality
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Participants will be divided into 2 groups: intervention and control groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive VR education program group (Experimental): Behavioral: Comprehensive VR Dementia Education Programviewed for cultural accuracy and adapted for Indonesian students.
  Interventions: Behavioral: Comprehensive VR Program
- Control Group (Active Comparator): Behavioral: Conventional Lecture Program
  Interventions: Behavioral: Conventional Lecture Program (Non-VR)

INTERVENTIONS:
Behavioral: Comprehensive VR Program — The intervention is a single-session VR dementia education program with up to 20 participants per session. The program includes: introduction; pre-program questionnaire; short lecture; bad drama video; a VR scenario showing poor communication; discussion; Lecture 1 on dementia; a positive VR scenario; good drama video; Lecture 2 on supporting people with dementia; N-impro activity; post-program questionnaire; and a brief conclusion. The program combines videos, VR experiences, lectures, and discussions to simulate real dementia care situations, build reflection, and strengthen students' knowledge, communication skills, and attitudes toward people living with dementia. All activities follow a fixed timeline to keep the session structured and ensure that each component supports the learning objectives. Content translated from Japanese will be reviewed for cultural accuracy and adapted for Indonesian students.
  Arms: Comprehensive VR education program group
Behavioral: Conventional Lecture Program (Non-VR) — The control group will receive a study explanation and complete the pre-test via Zoom. They will then follow a conventional dementia-related lecture program through the university's LMS, which includes lecture explanations, video lectures, and a discussion forum. Students will submit a written summary of the lecture as their assignment.
  After the LMS learning period ends, participants will attend a second Zoom session to complete the post-test.
  Arms: Control Group

SUMMARY:
This randomized controlled trial focuses on Indonesian nursing students and examines the effectiveness of virtual reality (VR) dementia education programs. The study addresses the following research questions:

1. What is the current level of knowledge and awareness about dementia among participants before they engage in a VR dementia education program?
2. What is the effect of a VR dementia education program on improving participants' attitudes, knowledge, and intention to help people living with dementia, and how satisfied are participants with the VR education program?

Participants will voluntarily join a 100-minute class session, with each participant attending only once. Participants are individually randomized into either the intervention group or the control group. The program is integrated into the faculty's dementia-related courses and includes several components: introduction, pre-program questionnaire, lecture, undesirable drama (unfriendly communication), undesirable VR experience, discussion, Lecture 1 (dementia overview), desirable VR experience, desirable drama, Lecture 2, N-impro, post-program questionnaire, and conclusion.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate a virtual reality (VR) dementia education program among nursing students in Indonesia. Participants will be nursing students enrolled in specific semesters and courses that have been selected for the implementation of this educational program. At Universitas Airlangga, the study will involve students in the fifth semester (third year). All prospective participants will be assigned new ID numbers to ensure confidentiality. This protocol has been reviewed and approved by the Ethics Committee of the Faculty of Nursing, Universitas Airlangga.

The VR dementia education program will be integrated into the Psychiatric Nursing course, which includes topics related to dementia care. Participants will be recruited during this course through in-class announcements. An overview of the study procedures will be provided, and detailed instructions will be given shortly before data collection begins. The research team will inform students about the study approximately one week in advance, and recruitment will take place via Google Forms. Students who agree to participate will receive their new ID numbers and details regarding the schedule and location of the program through class announcements three days before the intervention.

On the intervention day, participants will arrive at the designated location and sign the attendance list using their assigned IDs. The Principal Investigator (PI) will explain the study procedures and emphasize that participation is voluntary and that students may withdraw at any time without penalty. Students who choose not to participate will still receive standard dementia-related learning material through the university's e-learning platform, but they will not take part in the VR-based educational program. Students who agree to participate will provide informed consent and complete questionnaires before and after the intervention.

Eligible participants will be identified through the university's e-learning portal. Students registered in the selected courses for the 2025/2026 academic year will be screened at the beginning of the semester. All eligible students will receive comprehensive information about the study and an invitation to participate.

The research team will describe the study in person and distribute written information at the start of the course. The 2025/2026 course consists of four classes, each with approximately 50-60 students. All class will be randomly assigned to the intervention group. The intervention group will receive the comprehensive VR dementia education program, and the control group will receive standard dementia-related material via the e-learning platform. Both groups will complete pre- and post-intervention questionnaires. To evaluate long-term effects, follow-up data will be collected from both groups at the end of the course (expected February-March 2025).

The intervention group will participate in a single VR dementia education session, while the control group will receive a single standard lecture through the e-learning platform. Students who provide informed consent will complete the baseline survey (T1). In the intervention group, students will attend a classroom lecture and discussion on dementia (first class session) and then complete a post-lecture survey (T2). Both groups will then complete the final follow-up survey (T3) at the end of the semester. The control group will follow the same survey timeline (T1-T3).

ELIGIBILITY:
Inclusion Criteria:

* Nursing students enrolled in the designated semester at Universitas Airlangga.
* Students registered in the courses aligned with the implementation of the VR dementia education program.

Exclusion Criteria:

- Students who have prior experience with similar VR dementia education programs.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Attitudes Toward People Living with Dementia | - Baseline (before the intervention, on the same day as the session) - Immediately after the intervention (within 0-60 minutes after the session ends) - Long-term follow-up at 3 months after the intervention
  Participants' attitudes toward persons living with dementia (PLWD) will be assessed using the Attitudes Toward People with Dementia Scale, developed by Kim K and Kuroda K. (Kim K, Kuroda K. Factors related to attitudes toward people with dementia: Development of the Attitude Toward Dementia Scale and Dementia Knowledge Scale. Bulletin of Social Medicine. 2011; 28(1), 43-55). The original scale was published in Japanese, and a forward-backward translation process was conducted to produce the Indonesian version of the scale. The questionnaire consists of 14 items and is designed to assess participants' attitudes toward people with PLWD. The estimated time to complete the questionnaire is 3-5 minutes.

SECONDARY OUTCOMES:
Knowledge of Dementia | - Baseline (before the intervention, on the same day as the session) - Immediately after the intervention (within 0-60 minutes after the session ends) - Long-term follow-up at 3 months after the intervention
  Participants' knowledge of dementia will be assessed using the Dementia Knowledge Scale, developed by Kim and Kuroda (2011). This scale was originally designed to measure various aspects of dementia knowledge, including symptoms, causes, progression, and caregiving strategies. The scale consists of 15 multiple-choice and true/false questions that cover a broad range of dementia-related topics. The Indonesian version of the scale was created through a forward-backward translation process to ensure cultural and linguistic accuracy. Higher scores on this scale indicate a better understanding of dementia.
Intention to Help Persons Living with Dementia (PLWD) | - Baseline (before the intervention, on the same day as the session) - Immediately after the intervention (within 0-60 minutes after the session ends) - Long-term follow-up at 3 months after the intervention
  To assess participants' intention to help PLWD, we will use a set of four vignettes based on the study by Matsumoto et al. (2022). Each vignette presents a realistic scenario in which a person with dementia may need assistance, such as confusion in a public place, difficulty with daily tasks, or issues related to memory loss. Participants will read through each vignette and indicate their intended helping behavior on a 4-point Likert scale (ranging from "definitely would not help" to "definitely would help"). The vignettes are designed to assess the participants' willingness to offer practical, emotional, or social support to PLWD in everyday situations. The Indonesian version of the vignettes and Likert scale has also undergone a forward-backward translation to ensure that the language and context are appropriate for Indonesian nursing students.
Ageist Attitudes Towards Older Adults | - Baseline (before the intervention, on the same day as the session) - Immediately after the intervention (within 0-60 minutes after the session ends) - Long-term follow-up at 3 months after the intervention
  Participants' ageist attitudes will be assessed using selected items from the Fraboni Scale of Ageism (FSA). The FSA is a validated instrument developed by Fraboni et al. (1990) that measures stereotypes, prejudice, and discriminatory attitudes toward older adults. In this study, a subset of key items will be adapted and translated into Indonesian version using a forward-backward translation process to ensure cultural and linguistic appropriateness. The selected items cover three main domains: Stereotyping, Social distancing, Discriminatory attitudes. Each item will be rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree), with higher scores indicating stronger ageist attitudes. This measure will allow researchers to explore how underlying biases may impact students' empathy, communication, and willingness to provide equitable dementia care to older adults. This questionnaire is relevant to the study's aim of evaluating the impact of VR ASA not only on knowledg

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Airlangga, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
The IPD associated with participants' real IDs will be retained only by the PI of this study.
  New datasets will use new IDs so that only the PI can link the research data to participants' original IDs.
  Datasets that use the new IDs will be shared with the research team for data processing purposes (statistical analysis plan, SAP) and publication. All data will be stored for five years (Oktober 2024-Oktober 2029).
  Datasets will not be made public and will only be shared with the project's research team.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-11-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT07265856/Prot_SAP_ICF_000.pdf